CLINICAL TRIAL: NCT03655015
Title: Patient-derived Organoid Model and Circulating Tumor Cells for Treatment Response of Lung Cancer (CTMS 18-0056)
Brief Title: Patient-derived Organoid Model and Circulating Tumor Cells for Treatment Response of Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CTMS# 18-0056; HSC20180485H (Other: UT Health Science Center Institutional Review Board); R01CA269766 (NIH)
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Lung Neoplasm
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patient derived tumor specimens that are cultured into patient-derived organoids (PDOs)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Lung Tumor Resection — Lung Tumor Resection

SUMMARY:
Create a living biobank of PDOs from Stage I-III lung cancer patients.

DETAILED DESCRIPTION:
Creation a living biobank of PDOs from Stage I-IV lung cancer patients (n=50). We selected enrollment of at least 50 patients so that they can be risk stratified based on lung tumor type, staging and we plan to store these PDOs in biobank for future experiments. For each patient, tumor specimens will be collected at time of their surgery. No specific therapeutic intervention or treatment is provided as part of this study.

1. Establishment and culture of PDOs from lung cancer tumor specimens. PDOs will be biobanked for future experiments.
2. Lung organoids and CTCs will also be cultured and used to study baseline tumor characteristics using histology, immunohistochemistry, atomic force measurements; as well as, oncogenic signaling pathways and proteomic profile of lung organoids and CTCs derived from lung cancer patients (n>50).
3. Patient demographic information and data to be collected using a patient survey data sheet with treatment and survival history collected at pre-defined time period per the protocol schedule.

ELIGIBILITY:
Inclusion Criteria:

* Read, consented to and signed the IRB-approved informed consent form prior to any study related procedure.
* Diagnosis of lung cancer or lung mass or lymphadenopathy that will either systemic treatment or tumor resection as part of standard of care
* Any clinical stage of lung cancer
* Adult patients ≥18 years of age
* Able and willing to complete a questionnaire on their environmental/occupational exposures and smoking/alcohol history

Exclusion Criteria:

* At the discretion of the treating physician, patient will not be able to fulfill the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-10-16 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
To establish and characterize a biobank of patient-derived organoids (PDOs), and investigate the potential of PDOs to recapitulate ex vivo responses to chemotherapeutic and targeted agents observed in the clinic. | 10 years
  Establishment of a living biobank of PDOs and the potential of PDOs to repeat their process outside a living organism

SECONDARY OUTCOMES:
Correlation of PDO and Circulating tumor cells (CTCs) | 10 years
  To establish a connection between PDOs and CTCs, and their relationship to cancer

CONTACTS AND LOCATIONS:
Overall Officials: Josephine Taverna, MD, Principal Investigator — UT Health San Antonio M.D. Anderson Cancer Center
Locations (1):
- UT Health San Antonio, M.D. Anderson Cancer Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No